CLINICAL TRIAL: NCT05350995
Title: Evaluation of Antibiotherapy Prescribed for Outpatients From Emergency Departments
Acronym: EVAPAUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Clement OURGHANLIAN, Principal Investigator, Henri Mondor University Hospital
Other Study IDs: U2TI-001
Record Dates: First submitted 2022-03-15; First posted 2022-04-28 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Infectious Disease; Emergencies
MeSH Terms: conditions — Communicable Diseases; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
French health insurance data indicate that approximately 15% of ambulatory antibiotic consumption is generated by hospital prescriptions. This extra-hospital consumption represents a greater volume than intra-hospital consumption. To date, hospital indicators of good antibiotic use do not include this outpatient dimension. This study will provide a snapshot of the proportion of ambulatory antibiotics generated by emergencies and analyze compliance with management recommendations.This study will serve as a basis for developing indicators of outpatient antibiotic consumption generated by hospital activity and for identifying specific intervention targets aimed at the misuse situations that have been highlighted.

This study will be carried out in the form of a repeated survey on a given day (4 days, one across each season), carried out by the local mobile antibiotic therapy team, using a standardized grid. The survey will concern all the medical records of the patients visiting any emergency department on the days of the survey.

The evaluation of antibiotic therapies prescribed in discharge orders will be carried out in accordance with local management recommendations by the site investigator (infectious disease and/or emergency medicine specialist), who will assess whether the prescription is in accordance with the recommendations or not.

ELIGIBILITY:
Inclusion Criteria:

* Visit on emergency department on one of the survey days
* Age ≥18

Exclusion Criteria:

* Patient opposed to the collection of his/her data
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major outpatients visiting an emergency department on one of the survey days.
Sampling Method: Probability Sample
Enrollment: 9600 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Adequacy to local or national recommendations of antibiotic prescriptions identified on patient discharge prescriptions after a visit in emergency departments. | through study completion, an average of 1 year
  Adequacy to local or national recommendations (adequate/not adequate) of prescriptions, assessed by local investigator (infectious disease and/or emergency medicine specialist) at 4 days of collection: 1 day in each season (spring, summer, autumn and winter).

SECONDARY OUTCOMES:
Adequacy to the local or national recommendations of the antibiotic prescriptions identified on the patient discharge prescriptions by diagnosis. | Through study completion, an average of 1 year
  Adequacy to local or national recommendations (adequate/not adequate) of the antibiotic prescriptions identified on the patient discharge prescriptions by diagnosis assessed at 4 days of collection: 1 day in each season (spring, summer, autumn and winter).
Antibiotics prescription rate at discharge from emergency department. | Through study completion, an average of 1 year
Critical antibiotics prescription rate at discharge from emergency department. | Through study completion, an average of 1 year
  Critical antibiotics are defined by ANSM guidelines.
Factors associated with inadequacy to the local or national recommendations. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clément Ourghanlian, PharmD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- CHU Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No